CLINICAL TRIAL: NCT05401149
Title: Effectiveness and Safety of IV Rt-PA Treatment in Chinese AIS Patients Aged Above 80 Years: a Real-world Study
Brief Title: Alteplase Treatment in Elderly Acute Ischaemic Stroke (AIS) Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0135-0349
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IV rt-PA cohort: Acute Ischaemic Stroke (AIS) patients aged > 80 years who received intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) (Alteplase) within 4.5 hours of symptom onset
  Interventions: Drug: rt-PA
- Non-reperfusion cohort: Acute Ischaemic Stroke (AIS) patients aged > 80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive any reperfusion treatments

INTERVENTIONS:
Drug: rt-PA — Recombinant Tissue Plasminogen Activator
  Groups: IV rt-PA cohort

SUMMARY:
The objective of this study is to find out if Chinese Acute Ischaemic Stroke (AIS) patients older than 80 years benefit from intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) treatment within 4.5 hours of symptom onset in a real-world clinical setting.

ELIGIBILITY:
Inclusion criteria:

* Patients registered in the Zhejiang Stroke Quality Control Centre (ZSQCC) platform from Jan 2017 to Mar 2020
* > 80 years of age
* Diagnosed with AIS at admission
* Arrived or admitted to the hospital within 4.5 hours of symptom onset
* If treated with IV rt-PA: received IV rt-PA within 4.5 hours of symptom onset

Exclusion criteria:

* Documented Intravenous Thrombolysis (IVT) contraindication except age to IV rt-PA treatment according to the Summary of Product Characteristics (SmPC)
* Missing any one of the key data (age, gender, baseline National Institutes of Health Stroke Scale [NIHSS], time of symptom onset, time of hospital arrival or admission, IVT or not, time of IV rt-PA treatment)
* Received thrombolysis agents other than rt-PA (urokinase, tenecteplase, recombinant plasminogen activator, prourokinase, streptokinase)
* Received endovascular treatment
* Received IV rt-PA after 4.5 hours of symptom onset

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In this study, AIS patient data from 80 stroke centres in the Zhejiang Stroke Quality Control Centre (ZSQCC) platform from January 2017 to March 2020 will be used.
Sampling Method: Non-Probability Sample
Enrollment: 3058 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim (China) Investment Co., ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Yang J, Huang YH, Zhong W, Gong X, Chen Y, Chen Z, Jin H, Yan S, Huang L, Yuan CZ, Lou M. Effectiveness of intravenous recombinant plasminogen activator treatment in Chinese patients with acute ischaemic stroke aged over 80 years: a retrospective cohort study. Stroke Vasc Neurol. 2025 Apr 30:svn-2024-004004. doi: 10.1136/svn-2024-004004. Online ahead of print. PMID 40312065
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study (NIS) based on existing data collected from the Zhejiang Stroke Quality Control Centre (ZSQCC) platform of Acute Ischaemic Stroke (AIS) to compare the 1-year favourable neurological functional outcome of Chinese AIS patients aged > 80 years who received intravenous (IV) Recombinant Tissue Plasminogen Activator (rt-PA) treatment within 4.5 hours of symptom onset versus those who did not receive reperfusion therapy within 4.5 hours of symptom onset.
Pre-assignment Details: 98,330 AIS patients were registered in the ZSQCC platform from January 2017 to March 2020. Based on the protocol screening criteria, a total of 3058 patients were included in the final analysis. Then, the study cohorts (patients who received IV rt-PA and patients who did not receive reperfusion treatment) were matched 1:1 by baseline characteristics using the propensity score matching (PSM) method. Propensity score matched patients are 1560 patients.
Period: Overall Study
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Started (Propensity score matched patients) | 780 | 780
Completed | 780 | 780
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score matched (PSM) cohorts of AIS patients between the IV rt-PA and non-reperfusion groups (1:1). Patients >80 years old and registered in the Zhejiang Stroke Quality Control Centre (ZSQCC) platform from Jan 2017 to Mar 2020.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort | Total
Number analyzed (Participants) | 780 | 780 | 1560
Age, Continuous [Mean (Standard Deviation); unit: Years] | 85.2 (3.4) | 85.3 (3.7) | 85.2 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 413 | 396 | 809
  Male | 367 | 384 | 751
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Favourable Outcome (Modified Rankin Scale (mRS) 0-1) at 1 Year
Description: Percentage of patients with favourable outcome (modified Rankin Scale (mRS) 0-1) at 1 year.
  The modified Rankin Scale (mRS) is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, from 'perfect health without symptoms' to 'death'. 0 - No symptoms.
  1. - No significant disability.
  2. - Slight disability.
  3. - Moderate disability.
  4. - Moderately severe disability.
  5. - Severe disability.
  6. - Dead.
  Reported percentages of subjects were calculated from the conditional logistic regression models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline National Institutes of Health Stroke Scale (NIHSS) score, and time from symptom onset to hospital admission.
Time Frame: Up to 1 year post index hospital admission (between January 2017 and March 2020); data retrieved and studied from July 18, 2022 to December 14, 2022 (approximately 5 months of this study).
Population: Propensity score matched (PSM) cohorts of AIS patients between the IV rt-PA and non-reperfusion groups (1:1), clinical outcomes and baseline characteristics were compared between the matched cohorts. Patients >80 years old and registered in the Zhejiang Stroke Quality Control Centre (ZSQCC) platform from Jan 2017 to Mar 2020.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 780 | 780
Percentage of Participants | 27.7 [24.6 to 30.8] | 23.8 [20.9 to 26.8]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Odds Ratio (OR) (95% CI) and P values for this outcome were derived from the conditional logistic regression models with stratification by matching pairs and adjustment for prior modified Rankin Scale (mRS) score (≤ 1 or not), baseline National Institutes of Health Stroke Scale (NIHSS) score, and time from symptom onset to hospital admission; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.35 to 2.59] — IV rt-PA cohort/Non-reperfusion cohort

2. Secondary Outcome: Percentage of Patients With Any Intracranial Haemorrhage (ICH) During Hospitalisation
Description: Percentage of patients with any intracranial haemorrhage (ICH) during hospitalisation.
  Reported percentages of subjects were calculated from the conditional logistic regression models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline NIHSS score, and time from symptom onset to hospital admission.
Time Frame: Up to 3 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 780 | 780
Percentage of Participants | 13.7 [11.3 to 16.1] | 10.8 [8.6 to 12.9]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — OR (95% CI) and P values were derived from the conditional logistic regression models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline NIHSS score, and time from symptom onset to hospital admission; p = 0.054, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.99 to 2.06] — IV rt-PA cohort/Non-reperfusion cohort

3. Secondary Outcome: All-cause Mortality During Hospitalisation
Description: All-cause mortality during hospitalisation.
  Reported percentages of subjects were calculated from the conditional logistic regression models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline NIHSS score, and time from symptom onset to hospital admission.
Time Frame: Up to 3 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 780 | 780
Percentage of Participants | 4.5 [3.0 to 5.9] | 2.8 [1.7 to 4.0]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.097, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.88 to 4.86] — IV rt-PA cohort/Non-reperfusion cohort

4. Secondary Outcome: Percentage of Patients With Independence (Modified Rankin Scale (mRS) 0-2) at 1 Year
Description: Percentage of patients with independence (modified Rankin Scale (mRS) 0-2) at 1 year.
  The modified Rankin Scale (mRS) is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, from 'perfect health without symptoms' to 'death'. 0 - No symptoms.
  1. - No significant disability.
  2. - Slight disability.
  3. - Moderate disability.
  4. - Moderately severe disability.
  5. - Severe disability.
  6. - Dead.
  Reported percentages of subjects were calculated from the conditional logistic regression models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline National Institutes of Health Stroke Scale (NIHSS) score, and time from symptom onset to hospital admission.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 780 | 780
Percentage of Participants | 37.3 [33.9 to 40.7] | 33.7 [30.4 to 37.0]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.48 to 2.75] — IV rt-PA cohort/Non-reperfusion cohort

5. Secondary Outcome: Distribution of Modified Rankin Scale (mRS) Score at 1 Year
Description: Distribution of modified Rankin Scale (mRS) score at 1 year.
  The modified Rankin Scale (mRS) is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, from 'perfect health without symptoms' to 'death'. 0 - No symptoms.
  1. - No significant disability.
  2. - Slight disability.
  3. - Moderate disability.
  4. - Moderately severe disability.
  5. - Severe disability.
  6. - Dead.
  Reported percentages of subjects were calculated from the conditional logistic regression models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline National Institutes of Health Stroke Scale (NIHSS) score, and time from symptom onset to hospital admission.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 780 | 780
Units on a scale | 3.5 (2.4) | 3.7 (2.3)
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Odds Ratio (OR) (95% CI) and P values for this outcome were derived from the ordinal logistic regression models with adjustment for prior modified Rankin Scale (mRS) score (≤ 1 or not), baseline National Institutes of Health Stroke Scale (NIHSS) score, and time from symptom onset to hospital admission; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.64 to 0.93] — IV rt-PA cohort/Non-reperfusion cohort

6. Secondary Outcome: All-cause Mortality at 1 Year
Description: All-cause mortality at 1 year.
Time Frame: as for outcome 1
Population: Among PSM cohort (1560 patients), 120 patients (41 in IV rt-PA group; 79 in non-reperfusion therapy group) were excluded from the analysis due to missing date of death.
  To ensure that each matching pair has one patient from IV rt-PA group and one patient from non-reperfusion therapy group at the same time further 118 patients (78 in IV rt-PA group; 40 in non-reperfusion therapy group) were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
Number analyzed (Participants) | 661 | 661
Percentage of Participants | 36.2 [32.5 to 39.8] | 31.5 [27.9 to 35.0]
Statistical Analysis 1: Comparison: IV Rt-PA Cohort vs Non-reperfusion Cohort; Test type: Other — Hazard ratio (HR) (95% Confidence Interval) and P values were derived from the cox proportional hazards models with stratification by matching pairs and adjustment for prior mRS score (≤ 1 or not), baseline NIHSS score, and time from symptom onset to hospital admission; p = 0.077, Regression, Cox; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.98 to 1.64] — IV rt-PA cohort/Non-reperfusion cohort

ADVERSE EVENTS:
Time Frame: All-Cause-mortality: From the patient registration in the ZSQCC platform (between January 2017 and March 2020) to 1-year follow-up, up to 1 year.
Description: This is a non-interventional study (NIS) based on existing data from the Zhejiang Stroke Quality Control Centre (ZSQCC) platform. No adverse events were collected on an individual case level.
  Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
  All-Cause Mortality is an outcome of this study and thus additionally reported below.
Arm/Group | IV Rt-PA Cohort | Non-reperfusion Cohort
All-Cause Mortality (participants affected / at risk) | 308/780 | 303/780
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
According to Boehringer Ingelheim's internal policy, no document date is required in the title page of the Statistical and Epidemiological Analysis Plan

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT05401149/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT05401149/SAP_001.pdf